CLINICAL TRIAL: NCT04542785
Title: Lenient Rate Control Versus Strict Rate Control for Atrial Fibrillation. The Danish Atrial Fibrillation (DanAF) Randomised Clinical Trial
Brief Title: Lenient Rate Control Versus Strict Rate Control for Atrial Fibrillation. The Danish Atrial Fibrillation Randomised Clinical Trial
Acronym: DanAF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Holbaek Sygehus (Other)
Collaborators: Odense University Hospital (Other); Hvidovre University Hospital (Other); Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Joshua Rose-Hansen Feinberg, MD, Holbaek Sygehus
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REG-078-2019
Record Dates: First submitted 2020-08-26; First posted 2020-09-09 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Atrial Fibrillation, Persistent; Atrial Fibrillation Chronic; Atrial Fibrillation
Keywords: Rate control
MeSH Terms: conditions — Atrial Fibrillation | interventions — Heart Rate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Outcome assessors will be blinded. Participants will not be informed of the heart rate target or actual heart rate. Treatment providers managing the heart rate target will not be blinded as the intervention requires information of the heart rate. Other treatment providers will not be informed of the heart rate target.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lenient rate control (Experimental): Treating physicians will target a resting heart rate between 80 and 110 beats per minute on a 12-lead resting ECG measured over 1 minute after 5 minutes of rest.
  Interventions: Other: Rate control
- Strict rate control (Active Comparator): Treating physicians will target a resting heart rate a mean resting heart rate < 80 bpm on a 12-lead resting ECG measured over 1 minute after 5 minutes of rest.
  Interventions: Other: Rate control

INTERVENTIONS:
Other: Rate control — Treatment will be provided according to current guidelines and as such the algorithm for treatment will be differentiated based on the status of left ventricular ejection fraction. For participants with reduced left ventricular ejection fraction, beta-blockers (metoprolol and bisoprolol) will be the primary therapy. Secondary therapies may include digoxin or amiodarone. For participants with preserved left ventricular ejection fraction, the primary therapy will be beta-blockers (metoprolol and bisoprolol) or non-dihydropyridine calcium-channel blockers (verapamil) with secondary therapy consisting of digoxin or amiodarone. Pacing therapies, alone or with atrioventricular node ablation, are utilised as indicated in the view of the treating physician.

SUMMARY:
Atrial fibrillation is the most common heart arrhythmia with a prevalence of approximately 2% in the western world. Atrial fibrillation is associated with an increased risk of death and morbidity. The comparable effects of a lenient rate control strategy and a strict rate control strategy in patients with atrial fibrillation are uncertain and only one trial has assessed this previously in patients with permanent atrial fibrillation.

The investigators will therefore undertake a randomised, superiority trial at four hospitals in Denmark.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with atrial fibrillation (ECG confirmed and diagnosed by the treatment provider) who at inclusion have either persistent (defined as atrial fibrillation for more than 7days) or permanent atrial fibrillation (only rate control is considered going forward).
2. Rate control must be accepted as being the primary management strategy going forward. Consideration towards whether rhythm control is more appropriate must be considered, especially given the results of the Early treatment of Atrial fibrillation for Stroke prevention Trial (EAST).
3. Informed consent.
4. Adult (18 years or older).

Exclusion Criteria:

1. No informed consent.
2. Initial heart rate under 80 bpm at rest (assessed via ECG before randomisation).
3. Less than 3 weeks of anticoagulation with new oral anticoagulants or 4 weeks with efficient warfarin if indicated.
4. If the treating physician deems that the participant is not fit to be randomised into both groups based on an individual assessment. Such a decision will be made before randomisation by the treating physician. This can e.g. be participants dependent on a high ventricular rate to maintain a sufficient cardiac output. Such participants could be participants with heart failure, participants with a hemodynamically significant valve dysfunction, or severely dehydrated participants.
5. Participants who are haemodynamically unstable and therefore require immediate electrical cardioversion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2021-03-31 (Actual); Primary Completion 2026-03-02 (Estimated); Study Completion 2026-03-02 (Estimated)

PRIMARY OUTCOMES:
Short Form-36 (SF-36) physical component score | After 1 year

SECONDARY OUTCOMES:
Days alive outside hospital | After 6 months
Atrial Fibrillation Effect on Quality of Life (AFEQT) | After 1 year
Short Form-36 (SF-36) mental component score | 1 year
Serious adverse events | 1 year

OTHER OUTCOMES:
All-cause mortality | 1 year
  Mortality regardless of cause.
All-cause mortality | 2 year
  Mortality regardless of cause.
All-cause mortality | After 3 years
  Mortality regardless of cause.
Composite of all-cause mortality, stroke, myocardial infarction and cardiac arrest. | 1 year
Composite of all-cause mortality, stroke, myocardial infarction and cardiac arrest. | 2 year
Composite of all-cause mortality, stroke, myocardial infarction and cardiac arrest. | After 3 years
Cardiac mortality | 1 year
Cardiac mortality | 2 year
Cardiac mortality | After 3 years
Stroke | 1 year
  ICD-10 codes I60-I63.
Stroke | 2 year
  ICD-10 codes I60-I63.
Stroke | After 3 years
  ICD-10 codes I60-I63.
Hospitalisation for worsening of heart failure | 1 year
Hospitalisation for worsening of heart failure | 2 year
Hospitalisation for worsening of heart failure | After 3 years
Number of hospital admissions | 1 year
Number of hospital admissions | 2 year
Number of hospital admissions | After 3 years
Six-minute walking distance | 1 year
Six-minute walking distance | 2 year
Six-minute walking distance | After 3 years
Physical activity measured using a trial accelerometer or similar | 1 year
Physical activity measured using a trial accelerometer or similar | 2 year
Physical activity measured using a trial accelerometer or similar | After 3 years
Presence of sleep apnoea | 1 year
Presence of sleep apnoea | 2 year
Presence of sleep apnoea | After 3 years
Heart rate | 1 year
Heart rate | 2 year
Heart rate | After 3 years
Healthcare costs | 1 year
Healthcare costs | 2 year
Healthcare costs | After 3 years
Various biomarkers | 1 year
Various biomarkers | 2 year
Various biomarkers | After 3 years
Switch to rhythm control strategy | 1 year
Switch to rhythm control strategy | 2 year
Switch to rhythm control strategy | After 3 years
Implantation of a pacemaker or cardioverter-defibrillator | 1 year
Implantation of a pacemaker or cardioverter-defibrillator | 2 year
Implantation of a pacemaker or cardioverter-defibrillator | After 3 years
The questionnaire WorkQ | 1 year
The questionnaire WorkQ | 2 year
The questionnaire WorkQ | After 3 years
Echocardiography - Left ventricle dimensions | After 1 year
Echocardiography - Left ventricle dimensions | After 2 years
Echocardiography - Left ventricle dimensions | After 3 years
Echocardiography - systolic and diastolic function | After 1 year
Echocardiography - systolic and diastolic function | After 2 years
Echocardiography - systolic and diastolic function | After 3 years
Echocardiography - Right ventricle dimension | After 1 year
Echocardiography - Right ventricle dimension | After 2 years
Echocardiography - Right ventricle dimension | After 3 years
Echocardiography - Atrial dimensions | After 1 year
Echocardiography - Atrial dimensions | After 2 years
Echocardiography - Atrial dimensions | After 3 years
Echocardiography - pulmonary pressure | After 1 year
Echocardiography - pulmonary pressure | After 2 years
Echocardiography - pulmonary pressure | After 3 years
Short Form-36 (SF-36) physical component score | After 2 years
Short Form-36 (SF-36) physical component score | After 3 years
Days alive outside hospital | After 1 year
Days alive outside hospital | After 2 years
Days alive outside hospital | After 3 years
Atrial Fibrillation Effect on Quality of Life (AFEQT) | After 2 years
Atrial Fibrillation Effect on Quality of Life (AFEQT) | After 3 years
Short Form-36 (SF-36) mental component score | After 2 years
Short Form-36 (SF-36) mental component score | After 3 years
Serious adverse events | After 2 years
Serious adverse events | After 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Feinberg, MD, Principal Investigator — Holbaek University Hospital/University of Southern Denmark
Locations (4):
- Denmark (4):
  - Holbæk Hospital, Holbæk
  - Hvidovre University Hospital, Hvidovre
  - Odense University Hospital, Odense
  - Zealand University Hospital - Roskilde, Roskilde

IPD SHARING:
Plan to Share IPD: Yes
We will share anonymised data in a data repository.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Not possible to describe yet but will be made available within a timely manner after publication of results.
Access Criteria: Sharing will abide by the General Data Protection Regulation and the Danish data protections laws.

REFERENCES:
- [Derived] Cold IM, Feinberg JB, Brandes A, Davidsen U, Dixen U, Dominguez H, Gang UJO, Gluud C, Hadad R, Kristensen KE, van Le DT, Nielsen EE, Olsen MH, Pedersen OD, Raymond IE, Sajadieh A, Soja AMB, Jakobsen JC. Lenient rate control versus strict rate control for atrial fibrillation: a statistical analysis plan for the Danish Atrial Fibrillation (DanAF) randomized clinical trial. Trials. 2023 Apr 1;24(1):250. doi: 10.1186/s13063-023-07247-7. PMID 37005636
- [Derived] Feinberg JB, Olsen MH, Brandes A, Raymond L, Nielsen WB, Nielsen EE, Stensgaard-Hansen F, Dixen U, Pedersen OD, Gang UJO, Gluud C, Jakobsen JC. Lenient rate control versus strict rate control for atrial fibrillation: a protocol for the Danish Atrial Fibrillation (DanAF) randomised clinical trial. BMJ Open. 2021 Mar 31;11(3):e044744. doi: 10.1136/bmjopen-2020-044744. PMID 33789853